CLINICAL TRIAL: NCT00735306
Title: A Phase I/II Trial of Radiation, Avastin and Tarceva for Resectable or Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Phase I/II Trial of Radiation, Avastin and Tarceva for Pancreatic Adenocarcinoma
Acronym: TART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001597
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced; Unresectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Avastin, Tarceva and Radiation Therapy
  Interventions: Drug: Avastin; Drug: Tarceva; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Avastin — Avastin 10 mg/kg IV on days 1, 15 and 29 Begins the first day of radiation therapy
  Other Names: bevacizumab
Drug: Tarceva — Daily by mouth per assigned dose, for 5.5 weeks Begins the first day of radiation therapy
  Other Names: erlotinib
Radiation: Radiation Therapy — Radiation to the pancreas Monday through Friday for 28 treatments

SUMMARY:
The primary purpose of this trial is to define the maximum tolerated and/or recommended phase II dose of the combination of Avastin and Tarceva in patients undergoing radiation therapy for carcinoma of the pancreas. An additional primary objective is to describe the frequency and nature of grade III/IV and grade I/II toxicities associated with this regimen. Secondary objectives include describing 1-year disease-free survival and overall survival rates as well as to estimate clinical and pathologic complete response rates associated with this regimen.

DETAILED DESCRIPTION:
This is a phase I/II study in which up to 18 patients will be enrolled in the phase I portion and up to an additional 26 patients in the phase II portion. Patients will be treated with Tarceva (cohort specified dose), along with fixed doses of Avastin and radiation therapy.

Avastin will be given as an IV dose on days 1, 15, and 29. Tarceva will be given as a once daily by mouth. On radiation days Tarceva will be taken immediately before or after XRT.

XRT will be given to a total dose of 50.4 Gy in 28 fractions, each fraction given once daily on Monday through Friday for 5.5 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically and/or cytologically confirmed adenocarcinoma of the pancreas, T1-4, N0-1, M0. Patients should have disease for which combined modality therapy is indicated.
* Performance status 0-2
* Life expectancy > 3 months
* Adequate hematologic, renal, hepatic function
* Calculated creatinine Cl > 50 mL/min
* Use of effective means of contraception in patients of child-bearing potential.

Exclusion Criteria:

* No prior therapy for pancreatic cancer
* Previous treatment with bevacizumab or erlotinib
* Evidence of duodenal invasion or gastric outlet obstruction
* Presence of bleeding diathesis or coagulopathy
* History or prior arterial thrombotic event
* Conditions leading to inadequate gastrointestinal tract absorption
* Poorly controlled diarrhea .
* Presence of baseline proteinuria or renal dysfunction (CrCl < 50 (Cockcroft-Gault equation)
* Inadequately controlled hypertension
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Clinically significant peripheral vascular disease
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant or lactating females
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, or localized prostate cancer with a current PSA of <1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry.
* Comorbid conditions that would complicate safety or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czito, MD, Principal Investigator — Duke University Medical Center, Dept Radiation Oncology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiation: Avastin 10 mg/kg intravenous infusion day 1, 15 and 29 and Tarceva 100, 125 or 150 mg once daily by mouth and Radiation Therapy Mon-Fri for 28 treatments.
Period: Overall Study
Arm/Group | Chemoradiation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemoradiation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tarceva Maximum Tolerated Dose in mg
Description: Tarceva maximum tolerated dose in mg
Time Frame: 1 yr
Measure: Number; unit: mg
Arm/Group | Chemoradiation
Number analyzed (Participants) | 12
mg | 150

2. Secondary Outcome: Number of Dose Limiting Toxicities
Time Frame: Within 30 days of completing radiation
Measure: Number; unit: Events
Arm/Group | Chemoradiation
Number analyzed (Participants) | 12
Events | 0

3. Secondary Outcome: One Year Overall Survival From Time of Diagnosis
Description: One year survival from time of diagnosis for patients who completed this regimen
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Single Arm Avastin, Tarceva and Radiation Therapy: Avastin, Tarceva and Radiation Therapy
  Avastin: Avastin 10 mg/kg IV on days 1, 15 and 29 Begins the first day of radiation therapy
  Tarceva: Daily by mouth per assigned dose, for 5.5 weeks Begins the first day of radiation therapy
  Radiation Therapy: Radiation to the pancreas Monday through Friday for 28 treatments
Arm/Group | Single Arm Avastin, Tarceva and Radiation Therapy
Number analyzed (Participants) | 12
participants | 6

ADVERSE EVENTS:
Arm/Group | Chemoradiation
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation (N=12)
Anorexia (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 7 (7)
Hypertension (Vascular disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes